CLINICAL TRIAL: NCT00963443
Title: A Double Blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Acetylsalicylic Acid Combined With Pseudoephedrine, Compared With Acetylsalicylic Acid Alone, and Pseudoephedrine Alone, on Symptoms of Pain.
Brief Title: Acetylsalicylic Acid Combined With Pseudoephedrine in Common Cold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13700; 2009-011355-46 (EudraCT Number)
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Common Cold
Keywords: Aspirin Complex; Acetylsalicylic Acid; Pseudoephedrine; Common Cold
MeSH Terms: conditions — Common Cold | interventions — Aspirin; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465); Drug: Pseudoephedrine
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Arm 3 (Active Comparator)
  Interventions: Drug: Pseudoephedrine
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — 2 Sachets of 500 mg Aspirin Complex.
  Arms: Arm 1; Arm 2
Drug: Pseudoephedrine — 2 Sachets of 30 mg Pseudoephedrine
  Arms: Arm 1; Arm 3
Drug: Placebo — Matching Placebo
  Arms: Arm 4

SUMMARY:
The purpose of the study is to determine the effectiveness of an acetylsalicylic acid (aspirin) pseudoephedrine combination for the treatment of pain and congestion symptoms compared to the effectiveness of the individual components of the medicine and the placebo (dummy treatment that looks like the real thing).The combination product of acetylsalicylic acid / pseudoephedrine is already marketed in several European countries as Aspirin® Complex.

ELIGIBILITY:
Inclusion Criteria:

* Patient in general good health with suspected viral upper respiratory tract infection (common cold)

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduction of nasal congestion and relief of pain | 4 hours

SECONDARY OUTCOMES:
Area under the curve for nasal airflow conductance from baseline | 1h, 2h, 3h
Sum of subjective nasal congestion intensity differences | 1h, 2h, 3h, 4h and 1, 2, 3 days
Total subjective nasal congestion relief | 1h, 2h, 3h,4 h and 1, 2, 3 days
Global assessment of nasal congestion | 3 days
Global assessment of pain relief | 3 days
Sum of pain intensity differences | 1h, 2h, 3h, 4h and 1, 2, 3 days
Total pain relief | 1, 2, 3 days
Adverse Event collection and physical examination | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cardiff, South Glamorgan, United Kingdom

REFERENCES:
- See also: Click here and search for EMA Websynopsis results — http://www.clinicaltrialsregister.eu